CLINICAL TRIAL: NCT03284385
Title: A Phase 2 Study of AZD1775 in SETD2-Deficient Advanced Solid Tumor Malignancies
Brief Title: Testing AZD1775 in Advanced Solid Tumors That Have a Mutation Called SETD2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01670; NCI-2017-01670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10170 (Other: Yale University Cancer Center LAO); 10170 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Locally Advanced Clear Cell Renal Cell Carcinoma; Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Metastatic Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (adavosertib) (Experimental): Patients receive adavosertib PO QD on days 1-5 and 8-12. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775

SUMMARY:
This phase II trial studies how well adavosertib works in treating patients with SETD2-deficient solid tumors that have spread to other places in the body (advanced/metastatic). Adavosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria of adavosertib (AZD1775) in advanced solid tumor malignancies other than clear cell renal cell carcinoma with evidence of pathogenic loss of SETD2 using next-generation sequencing panel.

II. To determine the objective response rate by RECIST 1.1 criteria of AZD1775 in clear cell renal cell carcinoma with evidence of loss of SETD2 using next-generation sequencing panel.

SECONDARY OBJECTIVES:

I. To determine the clinical benefit rate and duration of response of AZD1775 in SETD2-deficient tumors other than clear cell renal cell carcinoma.

II. To determine the clinical benefit rate and duration of response of AZD1775 in SETD2-deficient clear cell renal cell carcinoma subgroup.

III. To characterize the safety profile of AZD1775. IV. To determine whether H3K36me3 expression by immunohistochemical assay is associated with clinical outcomes.

OUTLINE:

Patients receive adavosertib orally (PO) once daily (QD) on days 1-5 and 8-12. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Histologically confirmed locally advanced or metastatic solid tumor malignancy other than clear cell renal cell carcinoma with progression on at least one prior systemic therapy and presence of pathogenic loss of SETD2 detected in tumor tissue detected using a Clinical Laboratory Improvement Act (CLIA)-certified next generation sequencing panel (e.g. UCSF500, FoundationOne)
* Cohort B: Patients with histologically confirmed locally advanced or metastatic clear cell renal cell carcinoma (with clear cell component on pathology), who have been treated with at least one prior systemic therapy for locally advanced or metastatic disease, including either tyrosine kinase inhibitor and/or immune checkpoint inhibitor, with evidence of SETD2 mutation on CLIA-certified next generation sequencing panel

  * All next generation sequencing (NGS) sequencing reports will be reviewed by the University of California at San Francisco (UCSF) Molecular Tumor Board to verify pathogenicity of SETD2 mutation. Each NGS report will be redacted for Protected Health Information (PHI) prior to submission from investigational site to UCSF MTB.
* Measurable disease by RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin within normal institutional limits (WLN) or =< 1.5 x upper limit of normal (ULN) in patients with liver metastases; or total bilirubin =< 3 x ULN with direct bilirubin WLN in patients with well documented Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3.0 x institutional upper limit of normal (=< 5 x ULN if known liver metastases)
* Serum creatinine =< 1.5 x ULN, OR
* Creatinine clearance >= 45 ml/min (24 hour urine creatinine clearance or calculated by Cockcroft-Gault equation)
* Any prior radiation must have been completed at least 7 days prior to the start of study drugs, and patients must have recovered from any acute adverse effects prior to the start of study treatment
* Female patients who are not of child-bearing potential and fertile females of childbearing potential who agree to use adequate contraceptive measures from 2 weeks prior to the study and until 1 month after study treatment discontinuation, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 3 days prior to the start of study treatment
* Male patients willing to abstain or use barrier contraception (i.e. condoms) for the duration of the study and for 3 months after treatment stops
* Willingness and ability to comply with study and follow-up procedures
* Has read and understands the informed consent form and has given written informed consent prior to any study procedures

Exclusion Criteria:

* Use of anti-cancer treatment drug =< 21 days or 5 half-lives (whichever is shorter) prior to the first dose of AZD1775; for drugs for which 5 half-lives is =< 21 days, a minimum of 10 days between termination of the prior treatment and administration of AZD1775 treatment is required
* Previous radiation therapy completed =< 7 days prior to the start of study drugs
* Major surgical procedures =< 28 days of beginning study treatment, or minor surgical procedures =< 7 days; no waiting period required following port-a-cath or other central venous access placement
* Grade > 1 toxicity from prior therapy (except alopecia or anorexia)
* Patient has an inability to swallow oral medications; Note: patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN)
* No other anticancer-therapy (chemotherapy, immunotherapy, hormonal anti-cancer therapy, radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is to be permitted while the patient is receiving study medication; patients on luteinizing hormone-releasing hormone (LHRH) analogue treatment for more than 6 months are allowed entry into the study and may continue at the discretion of the investigator
* Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or hemorrhage for at least 2 weeks after treatment; must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrollment; patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Any known hypersensitivity or contraindication to the components of the study drug AZD1775
* Patient has had prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug; co-administration of aprepitant or fosaprepitant during this study is prohibited; the use of sensitive substrates of CYP3A4, such as atorvastatin, simvastatin and lovastatin, is also prohibited in this study; transporter studies (in vitro) have shown that AZD1775 is an inhibitor of breast cancer resistance protein (BCRP); herbal preparations are not allowed throughout the study; these herbal medications include but are not limited to: St. John's wort, kava, ephedra (ma hung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng; patients should stop using these herbal medications 7 days prior to first dose of study treatment
* Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) >= class 2

  * Unstable angina pectoris
  * Congestive heart failure
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
  * AZD1775 should not be given to patients who have a history of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected; AZD1775 has not been studied in patients with ventricular arrhythmias or recent myocardial infarction
* Mean resting corrected QT (QTc) interval using the Fridericia formula (QTcF) > 450 ms (i.e., grade 1 or higher) for males and > 470 ms for females on electrocardiogram (ECG) prior to initiation of study treatment obtained from 3 electrocardiograms (ECGs) obtained 2-5 minutes apart at study entry, or history of congenital long QT syndrome

  * If baseline QTc on screening ECG is > 450 ms for males or > 470 ms for females:

    * Check potassium and magnesium serum levels
    * Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm QTcF interval
  * For patients with baseline heart rate (HR) < 60 bpm or > 100 bpm, manual measurement of QT interval by cardiologist is required, with Fridericia correction applied to that manual measurement to determine the QTc for eligibility consideration
  * Note: For patients with HR 60-100 bpm, manual measurement of QTc interval is NOT required
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women; pregnant women are excluded from this study because AZD1775 is WEE1 inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD1775, breastfeeding should be discontinued if the mother is treated with AZD1775
* Prior treatment with WEE1 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. The median duration of response will be descriptively reported using Kaplan-Meier product limit method along with 95% confidence interval. The objective response rate between cohorts will be compared using the chi-squared test.

SECONDARY OUTCOMES:
Clinical benefit rate | Up to 2 years
  Will be defined as patients who experience either objective response or stable disease for >= 6 months from start of study treatment. The clinical benefit rate across the entire study cohort will be descriptively reported along with 95% confidence interval.
Duration of response | Up to 2 years
  The median duration of response will be descriptively reported using Kaplan-Meier product limit method along with 95% confidence interval.
Incidence and severity of adverse events | Up to 2 years
  Will be graded by Common Toxicity Criteria version 5.0, will be descriptively reported for the safety-evaluable population.
H3K36me3 mark | Up to 2 years
  Will be assessed by immunohistochemistry.
Progression free survival | Up to 2 years
  The median progression-free survival for each cohort will be determined using the Kaplan-Meier product limit method and compared between cohorts using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul R Aggarwal, Principal Investigator — Yale University Cancer Center LAO
Locations (29):
- United States (29):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Maldonado E, Rathmell WK, Shapiro GI, Takebe N, Rodon J, Mahalingam D, Trikalinos NA, Kalebasty AR, Parikh M, Boerner SA, Balido C, Krings G, Burns TF, Bergsland EK, Munster PN, Ashworth A, LoRusso P, Aggarwal RR. A Phase II Trial of the WEE1 Inhibitor Adavosertib in SETD2-Altered Advanced Solid Tumor Malignancies (NCI 10170). Cancer Res Commun. 2024 Jul 1;4(7):1793-1801. doi: 10.1158/2767-9764.CRC-24-0213. PMID 38920407